CLINICAL TRIAL: NCT01686724
Title: Efficacy of the Collaborative Life Skills Program
Brief Title: Study of the Collaborative Life Skills Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R324A120358
Record Dates: First submitted 2012-07-16; First posted 2012-09-18 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit Hyperactivity Disorder Symptoms
Keywords: Attention Deficit Hyperactivity Disorder; Psychosocial Intervention; Behavioral Intervention; School-home collaborative intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Commerce

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Business as Usual (BAU) (Other): This group receives services as usual in their schools. They will receive the intervention after follow-up measures are gathered.
  Interventions: Other: Business As Usual
- Collaborative Life Skills Intervention (CLS) (Experimental): CLS is a 12-week program and includes school, parent, and student components which are integrated via joint teacher, parent, and student meetings and use of integrated behavioral programs in the classroom, on the playground, and at home.
  Interventions: Behavioral: Collaborative Life Skills Intervention (CLS)

INTERVENTIONS:
Behavioral: Collaborative Life Skills Intervention (CLS) — CLS is a 12-week program and includes school, parent, and student components which are integrated via joint teacher, parent, and student meetings and use of integrated behavioral programs in the classroom, on the playground, and at home.
  Arms: Collaborative Life Skills Intervention (CLS)
Other: Business As Usual
  Arms: Business as Usual (BAU)

SUMMARY:
This study tests the effectiveness of a newly developed integrated school-home behavioral intervention for behaviors related to Attention Deficit Hyperactivity Disorder (ADHD). The intervention is implemented by school-based mental health professionals within school settings.

ELIGIBILITY:
Inclusion Criteria:

* Attending a participating school and in 2-5th grade
* Referral by LSP as a child with apparent ADHD-related problems
* ≥ 6 symptoms (item score ≥ 2) of Inattention or Hyperactivity-Impulsivity on the pooled parent and teacher Child Symptom Inventory
* ≥ 3 on the Impairment Rating Scale by parent and teacher (cross-situational impairment)
* FSIQ or VIQ ≥ 80 (necessary for cognitive demands of the child skills curriculum)
* Caretaker consents to participate in treatment, child assents to participate

Exclusion Criteria:

* Presence of conditions that are incompatible with this study's treatment.
* severe visual or hearing impairment,
* severe language delay,
* psychosis,
* pervasive developmental disorder
* Parent or child does not read or speak English or does not read or speak Spanish for our Spanish language implementation of CLS (inability to complete assessment measures or participate in group treatments).
* Child is in an all-day special education classroom (children in these classrooms are frequently receiving intensive behavior modification programs such that the intervention would be expected to require modification for use in these settings)
* Children taking psychotropic medication for any reason other than to treat ADHD
* Children planning to change (start or stop) psychotropic medication
* Children who have changed a regimen of psychotropic medication (started or stopped) within 30 days prior to screening

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 504 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of Attention Deficit Hyperactivity Disorder as defined by DSMIV/V. | change from baseline on ADHD symptoms at 12 weeks

SECONDARY OUTCOMES:
Homework Problems Checklist (HPC) | change from baseline in homework problems at 12 weeks
Academic Competency Evaluation Scale (ACES) | change from baseline in ACES at 12 weeks
Homework Problems Checklist (HPC) | change from baseline in homework problems at 7 months
Academic Competency Evaluation Scale (ACES) | change from baseline in ACES at 7 months
Children's Organizational Skills Scale (COSS) | change from baseline in COSS at 12 weeks
Children's Organizational Skills Scale (COSS) | change from baseline in COSS at 7 months
Observations of classroom/school behavior | change from baseline on observed on-task behavior at 12 weeks
Observations of classroom/school behavior | change from baseline in observed on-task behavior at 7 months
Academic achievement | change from baseline in academic achievement at 12 weeks
Academic Achievement | change from baseline in academic achievement at 7 months
Social Skills Improvement Scale | change from baseline in social/behavioral functioning at 12 weeks
Social Skills Improvement Scale | change from baseline in social/behavioral functioning at 7 months
Test of Life Skills Knowledge | change from baseline in life skills knowledge at 12 weeks
Test of Life Skills Knowledge | change from baseline in life skills knowledge at 7 months
Alabama Parenting Questionnaire | change from baseline in parenting practices at 12 weeks
Alabama Parenting Questionnaire | change from baseline in parenting practices at 7 months
Parenting Stress Index | change from baseline in parenting stress at 12 weeks
Parenting Stress Index | change from baseline in parenting stress at 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Pfiffner, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Pfiffner LJ, Rooney ME, Jiang Y, Haack LM, Beaulieu A, McBurnett K. Sustained Effects of Collaborative School-Home Intervention for Attention-Deficit/Hyperactivity Disorder Symptoms and Impairment. J Am Acad Child Adolesc Psychiatry. 2018 Apr;57(4):245-251. doi: 10.1016/j.jaac.2018.01.016. Epub 2018 Feb 8. PMID 29588050
- [Derived] Pfiffner LJ, Rooney M, Haack L, Villodas M, Delucchi K, McBurnett K. A Randomized Controlled Trial of a School-Implemented School-Home Intervention for Attention-Deficit/Hyperactivity Disorder Symptoms and Impairment. J Am Acad Child Adolesc Psychiatry. 2016 Sep;55(9):762-70. doi: 10.1016/j.jaac.2016.05.023. Epub 2016 Jul 1. PMID 27566117